CLINICAL TRIAL: NCT02890940
Title: Bridging the Gap: Using Video Art to Document the Human Face of Disease & Predict Quality of Life Assessments in Brain Tumor Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stefan Petranek, Associate Professor of Photography and Intermedia, Indiana University
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: 1604467360
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Brain Tumors; Quality of Life; Animal Assisted Therapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pet Therapy (Experimental)
  Interventions: Behavioral: Pet Therapy

INTERVENTIONS:
Behavioral: Pet Therapy — Patients will be asked to complete the standardized QLQ-C30/BN20 questionnaires. Following completion of the questionnaires, a trained pet therapy dog will be brought to the patients for approximately 10 minutes. After approximately 10 minutes, the dog will be removed and the patients will be asked to re-complete the standardized QLQ-C30/BN20 questionnaires. Patients will be photographed and videographed during this time.
  Finally, patients will be asked to talk about how their perspectives on life have changed with their diagnosis. These responses will be captured for use in the art exhibit created from images collected during the study.

SUMMARY:
The goal of this study is to explore whether facial expression changes in visual portraits correlate with Quality of Life (QOL) questionnaire responses before and after pet therapy sessions and to compare scores of QOL questionnaires before and after pet therapy.

DETAILED DESCRIPTION:
Through this pilot study, the investigators propose to create new intersections between video art and clinical care by photographing and videotaping patients with brain tumors before, during and after pet therapy sessions. This exploratory scholarship has two equally compelling goals. First, the artistic component of the project aims to create compelling slow motion video portraits of patients' willing to share their experiences of what it is like to confront such a grave illness. The goal is to put a human face on disease and share the endurance of the human spirit through art. Second, the scientific component will assess the potential of using facial video portraits as a novel and innovative way to measure Quality of Life (QOL) in lieu of questionnaires in brain tumor patients. In addition, the project will evaluate the effects of pet therapy on the QOL of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain tumors
* Willingness to participate in a brief pet therapy session with a dog
* Willingness to allow photographs, pictures and audio used in an art exhibit

Exclusion Criteria:

* Allergy to dogs
* Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Correlation of facial expression changes with QOL questionnaire responses | Immediately prior to therapy session to immediately after therapy session
  Will look to see if there is a correlation between facial expression changes in visual portraits with QOL questionnaire responses before and after pet therapy sessions

SECONDARY OUTCOMES:
Comparison of scores of QOL questionnaires before and after pet therapy | Immediately prior to therapy session to immediately after therapy session
  Will compare QOL questionnaire scores from before and after pet therapy sessions to see if there is a change after the pet therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mahua Dey, MD, Principal Investigator — Indiana University; Stefan Petranek, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Variations VII by John Cage (Experiments in Art & Technology), Artpix/Microcinema International, 2008, DVD.
- [Background] Jill Fox, Artists-In-Labs: Networking in the Margins (New York: SpringerWien, 2010)
- [Background] Karin Lipson, "Islip Exhibition Explores How Science Influences Art," The New York Times, October 22, 2015
- [Background] "The Scar Project," accessed January 12, 2016, http://www.thescarproject.org/
- [Background] "Ne Serait ce Qu' Une Seconde," The Mimi Foundation, accessed December 27, 2015. https://www.youtube.com/watch?v=GFVMe8w0Tx0.
- [Background] Ferry Q, Steinberg J, Webber C, FitzPatrick DR, Ponting CP, Zisserman A, Nellaker C. Diagnostically relevant facial gestalt information from ordinary photos. Elife. 2014 Jun 24;3:e02020. doi: 10.7554/eLife.02020. PMID 24963138
- [Background] Langner, O., Dotsch, R., Bijlstra, G., Wigboldus, D. H. J., Hawk, S. T., & van Knippenberg, A. (2010). Presentation and validation of the Radboud Faces Database. Cognition and Emotion, 24(8), 1377-1388.
- [Background] Taphoorn MJ, Sizoo EM, Bottomley A. Review on quality of life issues in patients with primary brain tumors. Oncologist. 2010;15(6):618-26. doi: 10.1634/theoncologist.2009-0291. Epub 2010 May 27. PMID 20507891
- [Background] Liu R, Page M, Solheim K, Fox S, Chang SM. Quality of life in adults with brain tumors: current knowledge and future directions. Neuro Oncol. 2009 Jun;11(3):330-9. doi: 10.1215/15228517-2008-093. Epub 2008 Nov 10. PMID 19001097